CLINICAL TRIAL: NCT03877068
Title: Management of Inpatient Hyperglycemia by Continuous Glucose Monitoring in Insulin-treated Patients With Diabetes: Dexcom G6 Intervention Study
Brief Title: Dexcom G6 Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IRB00107703
Record Dates: First submitted 2019-03-14; First posted 2019-03-15 (Actual); Results first posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus
Keywords: Glycemic control; Bedside point-of-care capillary glucose monitoring; Dexcom; Continuous glucose monitoring; Hyperglycemia; Inpatient
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Dexcom G6 CGM - Continues Glucose Monitoring sensor system (Experimental): Patients will wear a real-time Dexcom G6 CGM, which provide BG readings every 5 minutes for up to 10 days. In addition, patients will undergo POC testing before meals and bedtime per hospital protocol. Insulin therapy will be titrated based on daily CGM printouts, which will include BG readings, glycemic excursions, hypoglycemia and severe hyperglycemia values throughout the day. Patients will wear a CGM in the current approved insertion site, the abdomen, and in the upper arm.
  Interventions: Device: Dexcom G6 CGM - Continues Glucose Monitoring sensor system; Diagnostic Test: POC BG - Point-of-Care Blood Glucose monitoring
- POC BG - Point-of-Care Blood Glucose monitoring (Active Comparator): Glucose monitoring by POC testing will be performed before meals and at bedtime. Results will be uploaded in the electronic medical record (EMR) system. The research team together with the PCP team will adjust daily insulin orders based on POC readings (standard of care). In addition, patients will wear a 'blinded' CGM where no results will be visualized by patients, nursing staff, primary care physician (PCP) or research teams.
  Interventions: Diagnostic Test: POC BG - Point-of-Care Blood Glucose monitoring

INTERVENTIONS:
Device: Dexcom G6 CGM - Continues Glucose Monitoring sensor system — A blinded factory-calibrated continues glucose monitoring sensor system Dexcom G6 will be placed shortly after admission. Two CGM devices will be inserted in all patients - one in the abdomen and one in the arm to also assess differences in blood glucose readings between upper extremity and abdominal insertion sites. Information on CGM readings will be collected daily during the hospital stay up to 10 days using the Dexcom Studio software to download the Dexcom receiver data.
  Arms: Dexcom G6 CGM - Continues Glucose Monitoring sensor system
Diagnostic Test: POC BG - Point-of-Care Blood Glucose monitoring — Standard of care - bedside point-of-care (POC) capillary blood glucose (BG) monitoring will be done before meals and bedtime daily during the hospital stay up to 10 days.
  Other Names: Standard of Care capillary glucose test

SUMMARY:
The study will assess if Continuous Glucose Monitoring (CGM) represents a better tool to guide healthcare providers in adjusting insulin therapy, by providing a more complete 24-hour assessment of glucose values compared to Point of Care (POC) testing, during hospitalization and after hospital discharge in general medicine and surgery patients with Type 2 Diabetes (T2D) and Type 1 Diabetes (T1D).

DETAILED DESCRIPTION:
Diabetes is reported in 20-34% of hospitalized adult patients in general medicine and surgery units and there is a large body of literature showing a strong association between diabetes and increased hospital mortality and morbidity. Clinical guidelines have recommended the use of basal bolus insulin regimens as the preferred management approach of non-intensive care unit (ICU) patients with diabetes, as it has been shown to be effective in improving glycemic control and reducing hospital complications. However, hypoglycemia is a common adverse event of insulin therapy, with incidence rates ranging between 12% and 35% in randomized studies in non-ICU settings. The development of hypoglycemia, like hyperglycemia, has been associated with higher rates of hospital complications, higher health care resource utilization, and hospital mortality.

Bedside point-of-care (POC) capillary glucose monitoring is the standard of care to assess glycemic control in the hospital. Diabetes guidelines recommend bedside capillary POC testing before meals and at bedtime to assess glycemic control and to adjust insulin therapy in the hospital. In contrast to POC testing, continuous glucose monitoring (CGM) measures interstitial glucose every 5-15 minutes, thus providing a more complete glycemic profile during 24-hours compared to standard POC glucose testing. The study will assess if CGM represents a better tool to guide healthcare providers in adjusting insulin therapy by providing a more complete 24-hour assessment of glucose values compared to POC testing, during hospitalization and after hospital discharge in general medicine and surgery patients with T2D and T1D.

Participants will be randomized to have the standard of care POC testing plus wear a sham CGM or to wear a real-time Dexcom G6 CGM, which provide BG readings every 5 minutes for up to 10 days during hospitalization. At the point of hospital discharge, participants with poorly controlled diabetes will be invited to participate in an open label outpatient study where they will wear a Dexcom G6 CGM or sham device for 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years admitted to a general medicine or surgical services.
2. History of T1D or T2D receiving insulin therapy during hospital admission.
3. Subjects must have a randomization BG <400 mg/dL without laboratory evidence of diabetic ketoacidosis (bicarbonate < 18 milliequivalents per litre (mEq/L), potential of hydrogen (pH) < 7.30, or positive serum or urinary ketones).
4. Patients with expected hospital length-of-stay of 2 or more day

Exclusion Criteria:

1. Patients with acute illness admitted to the ICU or expected to require admission to the ICU.
2. Patients expected to require MRI procedures during hospitalization.
3. Patients with clinically relevant hepatic disease (diagnosed liver cirrhosis and portal hypertension), corticosteroid therapy, end-stage renal disease (dialysis), or anasarca (massive peripheral edema).
4. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
5. Female subjects who are pregnant or breast-feeding at time of enrollment into the study.
6. Coronavirus Disease 2019 (COVID-19) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital, Atlanta, Georgia
  - Grady Health System, Atlanta, Georgia
  - Univeristy of Maryland, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications for this study (including text, tables, figures, and appendices) will be available for sharing after de-identification.
Supporting Information: Study Protocol
Time Frame: Data will be available for sharing beginning 6 months after publication and ending 5 years after publication.
Access Criteria: Individual participant data will be made available for sharing with researchers who provide a methodologically sound proposals should email proposals to geumpie@emory.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Spanakis EK, Urrutia A, Galindo RJ, Vellanki P, Migdal AL, Davis G, Fayfman M, Idrees T, Pasquel FJ, Coronado WZ, Albury B, Moreno E, Singh LG, Marcano I, Lizama S, Gothong C, Munir K, Chesney C, Maguire R, Scott WH, Perez-Guzman MC, Cardona S, Peng L, Umpierrez GE. Continuous Glucose Monitoring-Guided Insulin Administration in Hospitalized Patients With Diabetes: A Randomized Clinical Trial. Diabetes Care. 2022 Oct 1;45(10):2369-2375. doi: 10.2337/dc22-0716. PMID 35984478
- [Derived] Spanakis EK, Singh LG, Siddiqui T, Sorkin JD, Notas G, Magee MF, Fink JC, Zhan M, Umpierrez GE. Association of glucose variability at the last day of hospitalization with 30-day readmission in adults with diabetes. BMJ Open Diabetes Res Care. 2020 May;8(1):e000990. doi: 10.1136/bmjdrc-2019-000990. PMID 32398351

RESULTS

PARTICIPANT FLOW:
Groups:
- Point-of-Care Blood Glucose Monitoring: Participants receiving blood glucose (BG) monitoring by point-of-care (POC) testing before meals and at bedtime during their hospital stay (up to 10 days). Results were uploaded in the electronic medical record (EMR) system. Daily insulin was adjusted based on POC readings, per standard of care. Participants wore a 'blinded' CGM, where no results were visualized by participants, nursing staff, primary care physicians or members of the research team.
- Dexcom G6 Continuous Glucose Monitoring (CGM) System: Participants wearing a real-time Dexcom G6 Continuous Glucose Monitoring (CGM), which provides blood glucose (BG) readings every 5 minutes during their hospital stay (up to 10 days). Participants also had point-of-care (POC) testing before meals and bedtime per hospital protocol. Insulin therapy was titrated based on daily CGM printouts, which included BG readings, glycemic excursions, hypoglycemia and severe hyperglycemia values throughout the day. Participants wore a CGM in the currently approved insertion sites of the abdomen and upper arm.
Period: Overall Study
Arm/Group | Point-of-Care Blood Glucose Monitoring | Dexcom G6 Continuous Glucose Monitoring (CGM) System
Started (Started inpatient portion of the study) | 94 | 91
Began Optional Outpatient Portion of Study | 52 | 53
Completed Optional Outpatient Portion of Study | 41 | 44
Completed (Completed inpatient portion of the study) | 85 | 88
Not Completed | 9 | 3
Not completed — Physician Decision | 9 | 3

BASELINE CHARACTERISTICS:
Population: The baseline analysis includes participants who completed the inpatient portion of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Point-of-Care Blood Glucose Monitoring | Dexcom G6 Continuous Glucose Monitoring (CGM) System | Total
Number analyzed (Participants) | 85 | 88 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.32 (9.50) | 57.24 (12.45) | 56.29 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 37 | 68
  Male | 54 | 51 | 105
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 58 | 57 | 115
  White | 19 | 24 | 43
  Hispanic | 6 | 6 | 12
  Other | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 85 | 88 | 173
Diabetes Type [Count of Participants; unit: Participants]
  Type 1 | 7 | 11 | 18
  Type 2 | 78 | 77 | 155

OUTCOME MEASURES:

1. Primary Outcome: Mean Daily Blood Glucose (BG) Concentration While Hospitalized
Description: A random (non-fasting) blood glucose measurement of 140 mg/dL or less is considered normal, while a measurement of 200 mg/dL or more indicates diabetes.
Time Frame: During hospitalization (up to 10 days)
Population: This analysis includes participants who were hospitalized for at least 24 hours. Six participants in the POC group and 5 participants in the Dexcom G6 CGM group were excluded as they stayed less than 24 hours in the hospital.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- POC Blood Glucose Monitoring: Participants receiving blood glucose (BG) monitoring by point-of-care (POC) testing before meals and at bedtime during their hospital stay (up to 10 days). Results were uploaded in the electronic medical record (EMR) system. Daily insulin was adjusted based on POC readings, per standard of care. Participants wore a 'blinded' CGM, where no results were visualized by participants, nursing staff, primary care physicians or members of the research team.
- Dexcom G6 CGM System: Participants wearing a real-time Dexcom G6 Continuous Glucose Monitoring (CGM), which provides blood glucose (BG) readings every 5 minutes during their hospital stay (up to 10 days). Participants also had point-of-care (POC) testing before meals and bedtime per hospital protocol. Insulin therapy was titrated based on daily CGM printouts, which included BG readings, glycemic excursions, hypoglycemia and severe hyperglycemia values throughout the day. Participants wore a CGM in the currently approved insertion sites of the abdomen and upper arm.
Arm/Group | POC Blood Glucose Monitoring | Dexcom G6 CGM System
Number analyzed (Participants) | 79 | 83
mg/dL | 186.8 (39) | 183.2 (40)

2. Primary Outcome: Percent of Time With BG Between 70-180 mg/dL While Hospitalized
Description: Glycemic control is measured by the percent of time with BG in the range of 70-180 mg/dL.
Time Frame: During hospitalization (up to 10 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time in range
Arm/Group | POC Blood Glucose Monitoring | Dexcom G6 CGM System
Number analyzed (Participants) | 79 | 83
percentage of time in range | 48.64 (24.25) | 54.51 (27.72)

3. Primary Outcome: Number of Clinically Significant Hypoglycemia Events While Hospitalized
Description: The mean number of clinically significant hypoglycemia events, defined as BG <54 mg/dl (3.0mmol/L), per participant is presented here.
Time Frame: During hospitalization (up to 10 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events per participant
Arm/Group | POC Blood Glucose Monitoring | Dexcom G6 CGM System
Number analyzed (Participants) | 79 | 83
events per participant | 0.56 (1.46) | 0.22 (0.59)

4. Secondary Outcome: Number of Hypoglycemia Events While Hospitalized
Description: The mean number of hypoglycemia events, defined as BG < 70 (<3.9 mmol/L), per participant during hospitalization is presented here.
Time Frame: During hospitalization (up to 10 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events per participant
Arm/Group | POC Blood Glucose Monitoring | Dexcom G6 CGM System
Number analyzed (Participants) | 79 | 83
events per participant | 1.15 (2.24) | 0.65 (1.26)

5. Secondary Outcome: Number of Nocturnal Hypoglycemia Events While Hospitalized
Description: The mean number of events of nocturnal hypoglycemia per participant are presented here. Nocturnal hypoglycemia occurs between the hours of 12:00 midnight and 6:00 ante meridiem (AM). Hypoglycemia is defined as BG < 70 mg/dL (<3.9 mmol/L) and severe hypoglycemia is defined as BG < 54 mg/dL (<3.0 mmol/L).
Time Frame: During hospitalization (up to 10 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events per participant
Arm/Group | POC Blood Glucose Monitoring | Dexcom G6 CGM System
Number analyzed (Participants) | 79 | 83
events per participant
  Hypoglycemia | 0.34 (0.83) | 0.20 (0.49)
  Severe hypoglycemia | 0.23 (0.72) | 0.08 (0.36)

6. Secondary Outcome: Percent of Time With Hypoglycemia While Hospitalized
Description: The percentage of time spent with BG below the desired range, during the day and night of hospitalization was assessed. Hypoglycemia is defined as BG < 70 mg/dL (<3.9 mmol/L) and severe hypoglycemia is defined as BG < 54 mg/dL (<3.0 mmol/L).
Time Frame: During hospitalization (up to 10 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time below range
Arm/Group | POC Blood Glucose Monitoring | Dexcom G6 CGM System
Number analyzed (Participants) | 79 | 83
percentage of time below range
  Hypoglycemia (BG < 70 mg/dL) | 2.15 (5.91) | 0.69 (2.15)
  Severe hypoglycemia (BG < 54 mg/dL) | 1.00 (3.74) | 0.32 (1.33)

7. Secondary Outcome: Percent of Time With Hyperglycemia While Hospitalized
Description: The percentage of time above the desired BG range, during the day and night while hospitalized was assessed.
Time Frame: During hospitalization (up to 10 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time above range
Arm/Group | POC Blood Glucose Monitoring | Dexcom G6 CGM System
Number analyzed (Participants) | 79 | 83
percentage of time above range
  BG > 180mg/dL | 49.21 (25.50) | 44.80 (27.89)
  BG > 250mg/dL | 17.08 (17.59) | 16.24 (19.63)

8. Secondary Outcome: Glycemic Variability Calculated by Mean Amplitude of Glycemic Excursions (MAGE) While Hospitalized
Description: Mean amplitude of glycemic excursions (MAGE), together with mean and standard deviation, is the parameter for assessing glycemic variability and is calculated based on the arithmetic mean of differences between consecutive peaks and nadirs of differences greater than one standard deviation of mean glycemia. It is designed to assess major glucose swings and exclude minor ones.
Time Frame: During hospitalization (up to 10 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | POC Blood Glucose Monitoring | Dexcom G6 CGM System
Number analyzed (Participants) | 79 | 83
mg/dL | 65.02 (39.10) | 61.24 (32.41)

9. Secondary Outcome: Differences in BG by CGM Devices Placed in the Abdomen and Upper Extremity While Hospitalized
Description: The mean absolute relative difference (MARD) reflects accuracy of the CGM glucose reading compared to the reference POC reading. This is the current standard for assessing accuracy of glucometer readings. Lower MARD indicates smaller differences between the CGM and meter value; a higher MARD value indicates larger differences. A three way and direct head-to-head comparison of data from the abdomen, upper arm and POC BG will be compared.
Time Frame: During hospitalization (up to 10 days)
Population: This analysis includes participants wearing a CGM device in the indicated bodily location.
Measure: Mean (Standard Deviation); unit: mg/dL
Units Other Than Participants: glucose readings
Arm/Group | Point-of-Care Blood Glucose Monitoring | Dexcom G6 Continuous Glucose Monitoring (CGM) System
Number analyzed (Participants) | 89 | 84
Number analyzed (glucose readings) | 1391 | 1345
mg/dL
  MARD CGM arm vs POC reading | 13.717 (11.720) | 12.771 (12.728)
  MARD CGM abdomen vs POC reading: number analyzed (Participants) | 79 | 83
  MARD CGM abdomen vs POC reading | 16.414 (13.778) | 15.670 (12.816)

10. Secondary Outcome: Number of Sensor Changes During Hospitalization
Description: Events related to sensor changes (blinded sensor for the POC group or real-time sensor for CGM group), such as removal for procedures or imaging, sensors failures, and sensors dislodgments were recorded.
Time Frame: During hospitalization (up to 10 days)
Population: as for outcome 1
Measure: Number; unit: count of sensor changes
Arm/Group | POC Blood Glucose Monitoring | Dexcom G6 CGM System
Number analyzed (Participants) | 79 | 83
count of sensor changes | 1 | 13

11. Secondary Outcome: Mean Daily BG Concentration After Discharge
Description: as for outcome 1
Time Frame: After hospital discharge (up to 10 days)
Population: This analysis includes participants who completed the outpatient portion of this study.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Point-of-Care Blood Glucose Monitoring | Dexcom G6 Continuous Glucose Monitoring (CGM) System
Number analyzed (Participants) | 41 | 44
mg/dL | 200.41 (55.94) | 199.65 (45.86)

12. Secondary Outcome: Percent of Time With BG Between 70-180 mg/dL After Discharge
Description: Glycemic control after hospital discharge is measured by the percent of time with BG in the range of 70-180 mg/dL.
Time Frame: After hospital discharge (up to 10 days)
Population: This analysis includes participants who completed the outpatient portion of this study.
Measure: Mean (Standard Deviation); unit: percentage of time in range
Arm/Group | Point-of-Care Blood Glucose Monitoring | Dexcom G6 Continuous Glucose Monitoring (CGM) System
Number analyzed (Participants) | 41 | 44
percentage of time in range | 43.42 (30.38) | 42.66 (26.34)

13. Secondary Outcome: Number of Clinically Significant Hypoglycemia Events After Discharge
Description: The mean number of clinically significant hypoglycemia events, defined as BG <54 mg/dl (3.0mmol/L), during the day and night after hospital discharge, per participant is presented here.
Time Frame: After hospital discharge (up to 10 days)
Population: This analysis includes participants who completed the outpatient portion of this study.
Measure: Mean (Standard Deviation); unit: events per participant
Arm/Group | Point-of-Care Blood Glucose Monitoring | Dexcom G6 Continuous Glucose Monitoring (CGM) System
Number analyzed (Participants) | 41 | 44
events per participant | 4.41 (6.28) | 2.30 (1.95)

14. Secondary Outcome: Number of Hypoglycemia Events After Discharge
Description: The mean number of hypoglycemia events, defined as BG < 70 (<3.9 mmol/L), per participant after hospital discharge is presented here.
Time Frame: After hospital discharge (up to 10 days)
Population: This analysis includes participants who completed the outpatient portion of this study.
Measure: Mean (Standard Deviation); unit: events per participant
Arm/Group | Point-of-Care Blood Glucose Monitoring | Dexcom G6 Continuous Glucose Monitoring (CGM) System
Number analyzed (Participants) | 41 | 44
events per participant | 5.20 (7.10) | 3.77 (3.73)

15. Secondary Outcome: Count of Participants With Hypoglycemia After Discharge
Description: Hypoglycemia is defined as BG < 70 mg/dL (<3.9 mmol/L) and severe hypoglycemia is defined as BG < 54 mg/dL (<3.0 mmol/L).
Time Frame: After hospital discharge (up to 10 days)
Population: This analysis includes participants who completed the outpatient portion of this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Point-of-Care Blood Glucose Monitoring | Dexcom G6 Continuous Glucose Monitoring (CGM) System
Number analyzed (Participants) | 41 | 44
Participants
  Hypoglycemia (BG < 70 mg/dL) | 37 | 42
  Severe hypoglycemia (BG < 54 mg/dL) | 36 | 38

16. Secondary Outcome: Percent of Time With Hyperglycemia After Discharge
Description: The percentage of time above the desired BG range, during the day and night after hospital discharge was assessed.
Time Frame: After hospital discharge (up to 10 days)
Population: This analysis includes participants who completed the outpatient portion of this study.
Measure: Mean (Standard Deviation); unit: percentage of time above range
Arm/Group | Point-of-Care Blood Glucose Monitoring | Dexcom G6 Continuous Glucose Monitoring (CGM) System
Number analyzed (Participants) | 41 | 44
percentage of time above range
  BG > 180mg/dL | 52.35 (30.57) | 54.96 (26.52)
  BG > 250mg/dL | 26.29 (27.31) | 23.03 (26.25)

17. Secondary Outcome: Glycemic Variability Calculated by Mean Amplitude of Glycemic Excursions (MAGE) After Discharge
Description: Mean amplitude of glycemic excursions (MAGE), together with mean and standard deviation, is the parameter for assessing glycemic variability and is calculated based on the arithmetic mean of differences between consecutive peaks and nadirs of differences greater than one standard of mean glycemia. It is designed to assess major glucose swings and exclude minor ones
Time Frame: After hospital discharge (up to 10 days)
Population: This analysis includes participants who completed the outpatient portion of this study.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Point-of-Care Blood Glucose Monitoring | Dexcom G6 Continuous Glucose Monitoring (CGM) System
Number analyzed (Participants) | 41 | 44
mg/dL | 58.55 (23.76) | 68.35 (46.68)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time consent to participate was given up to 10 days during hospitalization and up to 10 days after discharge (up to 20 days of monitoring).
Arm/Group | POC Blood Glucose Monitoring | Dexcom G6 CGM System
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/88
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/88
Other Adverse Events (participants affected / at risk) | 3/85 | 2/88
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | POC Blood Glucose Monitoring (N=85) | Dexcom G6 CGM System (N=88)
Minor bleeding with sensor insertion (Surgical and medical procedures) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT03877068/Prot_SAP_000.pdf